CLINICAL TRIAL: NCT05654766
Title: Development of a Method for Assessing the Functional Activity of Platelets for the Differential Diagnosis of Thrombocytopathies Using Flow Cytometry
Brief Title: Assesment of the Functional Activity of Platelets for the Differential Diagnosis of Thrombocytopathies
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Institute of Biophysics and Cell Engineering of National Academy of Sciences of Belarus (Other Government)
Collaborators: Belarusian Research Center for Pediatric Oncology, Hematology and Immunology (Other)
Responsible Party: Sponsor
Other Study IDs: IBCE_PL1
Record Dates: First submitted 2022-12-08; First posted 2022-12-16 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Immune Thrombocytopenia; Thrombocytopathy; Acute Leukemia; Hemorrhagic Disorders
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Blood Platelet Disorders; Hemorrhagic Disorders | interventions — Flow Cytometry; Platelet Aggregation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: Group of healthy adult and pediatric participants, whose blood platelets will be used to evaluate normal ranges of parameters in the flow cytometry PFT.
  Interventions: Diagnostic Test: Flow cytometry; Diagnostic Test: Platelet aggregation and plasma coagulation
- Hemorrhagic syndrome and Acute Leukemia: Group of pediatric participants with any manifestations of hemorrhagic syndrome and/or acute leukemia
  Interventions: Diagnostic Test: Flow cytometry; Diagnostic Test: Platelet aggregation and plasma coagulation

INTERVENTIONS:
Diagnostic Test: Flow cytometry — Parameters such as FSC, SSC, median fluorescence of anti CD42b, PAC-1, CD41, CD63, CD62P, as well as Annexin V fluorescence will be assessed.
Diagnostic Test: Platelet aggregation and plasma coagulation — Turbodimetric platelet aggregation test, impedance platelet aggregation test. Standard plasma coagulation test (fibrinogen level, prothrombin test, thrombin time, activated partial thromboplastin time (aPTT)).

SUMMARY:
The purpose of this study is to develop a highly sensitive method for assessing the functional activity of platelets for use in the differential diagnosis of thrombocytopenia and platelet defects.

DETAILED DESCRIPTION:
The purpose of this study is to develop a highly sensitive method for assessing the functional activity of platelets using flow cytometry and turbidimetric and impedance aggregometry for use in the differential diagnosis of thrombocytopenia and platelet defects

ELIGIBILITY:
Inclusion Criteria:

* Pediatric participants with hemorrhagic syndrome (hemorrhagic rash, bruising, bleeding, increased bleeding of the skin and mucous membranes, spontaneous hemorrhages in soft tissues and joints)
* Pediatric participants with acute leukemia
* Parameters of the plasma level of blood coagulation correspond to the age normal levels

Exclusion Criteria:

* Anticoagulation drug therapy
* Antiaggregation drug therapy
* Biologically active additives

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy pediatric volunteers aged 1 to 17. Pediatric volunteers aged 1 to 17 with any manifestation of hemorrhagic syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-01-02 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Expression of CD42b by platelets | baseline
  Assessment of platelet functional activity by the detection of CD42b
Expression of CD41 by platelets | baseline
  Assessment of platelet functional activity by the detection of CD41
Expression of PAC-1 by platelets | baseline
  Assessment of platelet functional activity by the detection of PAC-1
Expression of CD63 by platelets | baseline
  Assessment of platelet functional activity by the detection of CD63
Expression of CD62p by platelets | baseline
  Assessment of platelet functional activity by the detection of CD62p
Expression of Annexin V by platelets | baseline
  Assessment of platelet functional activity by the detection of Annexin V
Level of platelet aggregation | baseline
  Assessment of platelet functional activity by turbidimetric aggregometry
Impedance of platelet aggregates | baseline
  Assessment of platelet functional activity by impedance aggregometry
Fibrinogen level | baseline
  Assessment of blood coagulation using Fibrinogen level test
Prothrombin test | baseline
  Assessment of blood coagulation using Prothrombin test
Thrombin time | baseline
  Assessment of blood coagulation using Thrombin time test
aPTT | baseline
  Assessment of blood coagulation using aPTT

CONTACTS AND LOCATIONS:
Overall Officials: rrchypp@gmail.com Shamova, Dr, Study Director — the Institute of Biophysics and Cell Engineering of National Academy of Sciences of Belarus; Viacheslav Dmitriev, Dr, Study Director — Belarussian Research Center for Pediatric Oncology, Hematology and Immunology

IPD SHARING:
Plan to Share IPD: No